CLINICAL TRIAL: NCT02846610
Title: Improvement of Acute Pain Treatment With Systemic and Regional Anesthesia
Brief Title: Registry for Acute Pain Treatment
Status: Terminated | Type: Observational
Why Stopped: The registry has a new setpup and a new entry
Sponsor: University Hospital, Saarland (Other)
Collaborators: Charite University, Berlin, Germany (Other); Ruhr University of Bochum (Other); HELIOS Hospital, Bad Saarow, Germany (Unknown); Technische Universität Dresden (Other); HELIOS Hospital, Erfurt, Germany (Other); Goethe University (Other); BG Unfallklinik Frankfurt am Main (Network); University of Hamburg-Eppendorf (Other); Diakoniekrankenhaus Friederikenstift (Other); Jena University Hospital (Other); Hospital Ludwigsburg, Germany (Unknown); Philipps University Marburg (Other); Hospital Memmingen, Germany (Unknown); St. Marien-Krankenhaus, Siegen, Germany (Unknown); Städtisches Klinikum gGmbH, Solingen, Germany (Unknown); University Hospital Freiburg (Other); University Hospital Muenster (Other); University Hospital of Cologne (Other); HELIOS Klinikum Lengerich (Unknown); Berlin DRK Hospital (Unknown); Diakonie Hospital Bad Kreuznach (Unknown); Ev. Hospital Unna (Unknown); Josephs Hospital Warendorf (Unknown); University Hospital Ulm (Other); Johannes Gutenberg University Mainz (Other)
Responsible Party: Sponsor
Organization: Universität des Saarlandes (Other)
Other Study IDs: NRA
Record Dates: First submitted 2016-05-28; First posted 2016-07-27 (Estimated); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Pain, Postoperative; Regional Anesthesia
Keywords: anesthesia; continuous regional anesthesia; complications; epidural analgesia; antibiotics
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- regional anesthesia: surgical patients (age: 0-100 years) having regional anesthesia along with the procedure and postoperative course
- systemic analgesia: surgical patients (age: 0-100 years) having systemic analgesia along with the procedure and post procedure course

SUMMARY:
The German Network for acute pain management and Regional Anesthesia (NRA) is a multi-center, non-interventional registry and benchmark project, assessing and analysing clinical and patient-reported procedural and outcome data of systemic analgesia and regional anesthesia hosted by the German Society of Anesthesia and Intensive Care Medicine (DGAI) and professional Society German Anesthetists (BDA)

DETAILED DESCRIPTION:
NRA offers the systematic documentation of patient related and procedure related components for acute pain treatments during and after surgery.

NRA collects preoperative, intraoperative, and postoperative data from treating physicians who complete a standard form. Data are collected concurrently with patient care by pain nurses or treating physicians and include detailed information about the medical conditions of patients having acute pain treatment along with the procedure and postoperative course.

The registry provides the basis for large scale analyses and benchmarks for several parameters.

The registry also aims at performing population-based research. Furthermore, its infrastructure allows for the conduct of prospective studies comparing the effectiveness of processes of care.

ELIGIBILITY:
Inclusion Criteria:

* The investigators include anonymous data from patients with continuous regional anesthesia, single shot regional anesthesia, or systemic analgesia

Exclusion Criteria:

* None.

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Surgical and non-surgical patients with continuous regional anesthesia, single shot regional anesthesia, or intravenous patient-controlled analgesia
Sampling Method: Probability Sample
Enrollment: 224744 (Actual)
Dates: Start 2007-09; Primary Completion 2023-05-11 (Actual); Study Completion 2023-05-11 (Actual)

PRIMARY OUTCOMES:
Acute complications during insertion of regional anesthesia | at the day of insertion, day zero
  Procedural complications include dural puncture, bleeding, nerve damage, intoxication, malfunction, technical and equipment difficulties or failures.

SECONDARY OUTCOMES:
Pain levels after surgery | Daily visits (ward rounds) as long as in-hospital pain treatment is given; may take up to the length of the hospital stay, up to 90 days
  Pain and pain related outcome measures (NRS at rest and on exertion, opioid and non-opioid consumption), interference of pain with activities, pain therapy side effects, pre-hospital existence of pain, information on general treatment
Satisfaction | after end of acute pain treatment, between day zero and up to day 90
  1. Patient and physician satisfaction: Satisfaction with the respective pain treatment reported by patients (verbal numeric rating scale ranging from 0 (=completely dissatisfied) to 10 (=completely satisfied).
Complications of acute pain treatment | Daily visits (ward rounds) as long as in-hospital pain treatment is given; may take up to the length of the hospital stay, between day zero and day 90
  hypotension, sedation, urinary retention, infections, procedural complications such as nausea and vomiting, respiratory depression, itching, malfunction, nerve damage, intoxication, technical and equipment difficulties or failures

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Volk, MD, Study Director — University Hospital, Saarland
Locations (1):
- Saarland University Medical Center, Homburg, Saarland, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Volk T, Engelhardt L, Spies C, Steinfeldt T, Kutter B, Heller A, Werner C, Heid F, Burkle H, Koch T, Vicent O, Geiger P, Kessler P, Wulf H. [A German network for regional anaesthesia of the scientific working group regional anaesthesia within DGAI and BDA]. Anasthesiol Intensivmed Notfallmed Schmerzther. 2009 Nov;44(11-12):778-80. doi: 10.1055/s-0029-1242127. Epub 2009 Nov 16. German. PMID 19918710
- [Background] Bomberg H, Kubulus C, Herberger S, Wagenpfeil S, Kessler P, Steinfeldt T, Standl T, Gottschalk A, Stork J, Meissner W, Birnbaum J, Koch T, Sessler DI, Volk T, Raddatz A. Tunnelling of thoracic epidural catheters is associated with fewer catheter-related infections: a retrospective registry analysis. Br J Anaesth. 2016 Apr;116(4):546-53. doi: 10.1093/bja/aew026. PMID 26994232
- [Background] Bomberg H, Albert N, Schmitt K, Graber S, Kessler P, Steinfeldt T, Hering W, Gottschalk A, Standl T, Stork J, Meissner W, Tessmann R, Geiger P, Koch T, Spies CD, Volk T, Kubulus C. Obesity in regional anesthesia--a risk factor for peripheral catheter-related infections. Acta Anaesthesiol Scand. 2015 Sep;59(8):1038-48. doi: 10.1111/aas.12548. Epub 2015 Jun 4. PMID 26040788
- [Background] Bomberg H, Kubulus C, List F, Albert N, Schmitt K, Graber S, Kessler P, Steinfeldt T, Standl T, Gottschalk A, Wirtz SP, Burgard G, Geiger P, Spies CD, Volk T; German Network for Regional Anaesthesia Investigators. Diabetes: a risk factor for catheter-associated infections. Reg Anesth Pain Med. 2015 Jan-Feb;40(1):16-21. doi: 10.1097/AAP.0000000000000196. PMID 25474624
- [Background] Volk T, Engelhardt L, Spies C, Steinfeldt T, Gruenewald D, Kutter B, Heller A, Werner C, Heid F, Burkle H, Gastmeier P, Wernecke KD, Koch T, Vicent O, Geiger P, Wulf H. [Incidence of infection from catheter procedures for regional anesthesia: first results from the network of DGAI and BDA]. Anaesthesist. 2009 Nov;58(11):1107-12. doi: 10.1007/s00101-009-1636-7. German. PMID 19890612
- [Background] Kubulus C, Schmitt K, Albert N, Raddatz A, Graber S, Kessler P, Steinfeldt T, Standl T, Gottschalk A, Meissner W, Wirtz SP, Birnbaum J, Stork J, Volk T, Bomberg H. Awake, sedated or anaesthetised for regional anaesthesia block placements?: A retrospective registry analysis of acute complications and patient satisfaction in adults. Eur J Anaesthesiol. 2016 Oct;33(10):715-24. doi: 10.1097/EJA.0000000000000495. PMID 27355866
- [Derived] Bomberg H, Huth A, Wagenpfeil S, Kessler P, Wulf H, Standl T, Gottschalk A, Doffert J, Hering W, Birnbaum J, Spies C, Kutter B, Winckelmann J, Burgard G, Vicent O, Koch T, Sessler DI, Volk T, Raddatz A. Psoas Versus Femoral Blocks: A Registry Analysis of Risks and Benefits. Reg Anesth Pain Med. 2017 Nov/Dec;42(6):719-724. doi: 10.1097/AAP.0000000000000643. PMID 28806216